CLINICAL TRIAL: NCT01478035
Title: Efficacy of Phenytoin in the Prophylaxis of Seizures of Patients With Pneumococcal Meningitis at Least 50 Yrs Old. A Multi-center Comparative Randomized Double-blind and Placebo-controlled Clinical Trial
Brief Title: Study on the Efficacy of Phenytoin in the Prophylaxis of Seizures of Patients With Pneumococcal Meningitis at Least 50 Yrs Old.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: M. Carmen Cabellos Minguez (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Hospital Vall d'Hebron (Other); Germans Trias i Pujol Hospital (Other); Hospital Clinic of Barcelona (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Juan Canalejo (Other); Hospital Mutua de Terrassa (Other); Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor-Investigator, M. Carmen Cabellos Minguez, Medical Doctor, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INFSNC1
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Seizures; Pneumococcal Meningitis
Keywords: Phenytoin prophylaxis; Pneumococcal meningitis; Randomized; Placebo-controlled; Double blind; Patient 50 years or older
MeSH Terms: conditions — Seizures; Meningitis, Pneumococcal | interventions — Phenytoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phenytoin prophylaxis (Experimental): Patients with suspected or proven pneumococcal meningitis are allocated to receive phenytoin prophylaxis or placebo to avoid seizures during the 10 days of antibiotic therapy starting after the antibiotic therapy
  Interventions: Drug: Phenytoin
- placebo (Placebo Comparator): placebo vials and pills labeled as phenytoin prophylaxis vials and pills
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Phenytoin — Phenytoin 18 mg /Kg/day iv as loading dose. 24 hours later phenytoin 6 mg/Kg/d in 3 divided doses iv shifting to oral route at the same dose when the patient is able to use oral route.
  Arms: phenytoin prophylaxis
Drug: placebo — Placebo 18 mg /Kg/day iv as loading dose. 24 hours later placebo 6 mg/Kg/d in 3 divided doses iv shifting to oral route at the same dose when the patient is able to use oral route.
  Arms: placebo

SUMMARY:
To evaluate the efficacy of the prophylaxis with phenytoin in the prevention of seizures in patients with pneumococcal meningitis. Hypothesis: Administration of prophylactic phenytoin will reduce the incidence of seizures in patients with pneumococcal meningitis older than 50 yrs.

DETAILED DESCRIPTION:
Background: Bacterial meningitis has still a high morbi-mortality despite the global improvement in therapy.

Among complications, the presence of seizures may contribute to increase the morbi-mortality. Prophylactic phenytoin is used in clinical practice in high risk patients but this use is variable because there are not controlled clinical trials demonstrating efficacy along with antibiotics and corticosteorids. Pneumococcal episodes are associated to a higher number of seizures and a higher mortality especially in elderly patients.

Objectives: To evaluate the efficacy of the prophylaxis with phenytoin in the prevention of seizures in patients with pneumococcal meningitis. Hypothesis: Administration of prophylactic phenytoin will reduce the incidence of seizures in patients with pneumococcal meningitis older than 50 yrs.

Methodology: Multicentre, randomized, double blind placebo controlled clinical trial. Patients will be included mostly from hospitals from REIPI and CAIBER and randomly assigned to receive phenytoin or placebo.

Sample size has been estimated in 61 patients per group. Antibiotic therapy and ICP prophylaxis will be standardized in all centres. Phenytoin administration will be maintained during antibiotic therapy. End point will be incidence of seizures during hospital stay and overall mortality will be a secondary end-point. Followup visits at 1 and 3 month will be performed.

ELIGIBILITY:
Inclusion Criteria:

Adult patients > or = 50 years old.

Diagnosed of pneumococcal meningitis due to clinical characteristics plus a positive CSF Gram stain and/or a detection of pneumococcal antigen or PCR

or

Suspected pneumococcal meningitis since it is an episode related to otitis, pneumonia, sinusitis or pericranial fistula or in patients with known risk factors such as myeloma or splenectomy.

Exclusion Criteria:

To have seizures prior to arrive to the hospital or the inclusion in the study.

Pregnancy or breastfeeding.

To have conduction abnormalities in ECG.

History of allergy or intolerance to phenytoin.

Patients with meningitis as a complication of neurosurgical procedures.

Epileptic patients taking usually anticonvulsivants.

Refusal by the patient or family to participate and/or to sign the informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Presence of seizures (clinical) after initiation of phenytoin /placebo prophylaxis during the 10 days of antibiotic therapy | 10 days
  Presence of seizures (clinical) after initiation of phenytoin /placebo prophylaxis during the 10 days of antibiotic therapy

SECONDARY OUTCOMES:
Need for anticonvulsivant therapy at 3 months | 3 months
  Need for anticonvulsivant therapy at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Carmen Cabellos, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (4):
- Spain (4):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Juan Canalejo, A Coruña
  - Fundacio Institut per la Recerca de l'hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Virgen del Rocio, Seville